CLINICAL TRIAL: NCT02760472
Title: A Randomised Intervention Single Center Study to Determine the Role of Fatty Acids in Serum in Preventing Retinopathy of Prematurity
Brief Title: A Fatty Acids Study in Preventing Retinopathy of Prematurity
Acronym: DonnaMega
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Carola Pfeiffer-Mosesson (Other)
Responsible Party: Sponsor-Investigator, Carola Pfeiffer-Mosesson, Research Nurse, Queen Silvia Children's Hospital, Gothenburg, Sweden
Organization: Queen Silvia Children's Hospital, Gothenburg, Sweden (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2008-000046-31
Record Dates: First submitted 2016-03-30; First posted 2016-05-03 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Retinopathy of Prematurity
Keywords: Retinopathy of Prematurity; Preterm; Fatty acids
MeSH Terms: conditions — Retinopathy of Prematurity; Premature Birth | interventions — SMOFlipid; ClinOleic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinoleic (Active Comparator): Parenteral fatty acid supplementation to preterm infants in preventing retinopathy of prematurity
  Interventions: Drug: Clinoleic
- SMOFlipid (Experimental): Parenteral fatty acid supplementation to preterm infants in preventing retinopathy of prematurity
  Interventions: Drug: SMOFlipid

INTERVENTIONS:
Drug: SMOFlipid — Parenteral fatty acid supplementation to preterm infants in preventing retinopathy of prematurity
  Arms: SMOFlipid
Drug: Clinoleic — Parenteral fatty acid supplementation to preterm infants in preventing retinopathy of prematurity
  Arms: Clinoleic

SUMMARY:
Most fatty acids, important for development and especially the Omega-3 fatty acids for the brain development are transferred in the third trimester with means that in the premature infant this transport via the placenta is interrupted and the infant is dependent on the concentrations in breast milk which vary depending on the mother's diet and her stores. It has even been suggested that low Omega-3 would be a cause of premature delivery. Many countries have much higher levels of Omega-3 fatty acids in breast milk than found in Sweden and breast milk substitutions are generally now supplemented with the Long Chained Poly Unsaturated Fatty Acids (LCPUFA). Therefore the supplementation to be given can not be seen to give any risks for the infant. On the contrary, several studies have shown that mother who eat equal to or less than twice fish a week during pregnancy give birth to infants with impaired development.

Low Omega-3 levels in premature infants between gestational ages of 23 and 40 weeks can be one reason for Retinopathy of Prematurity (ROP) development. Restoration of Omega-3, Dokosahexaenacid (DHA) and Eikosapentaenacid (EPA) to normal in utero levels may prevent ROP by allowing normal vessel growth and survival. An increase of Omega-3 levels bringing levels to within physiological range may prevent development of ROP.

DETAILED DESCRIPTION:
The study is a Randomised Intervention, Single-Center Study to Determine the Role of Fatty Acids in Serum and Breast Milk in preventing Retinopathy of Prematurity.

Subjects who meet all inclusion and none of the exclusion criteria will be enrolled into the study. Upon entry into the study, subjects will be randomized and given a unique subject number.

A randomised intervention study of 45+45 infants without major malformations born with a gestational age less than 28 weeks + 0 days will be performed.

Randomization of the patients to either:

1. Conventional fatty acid supplementation regime with Clinoleic (with Vitalipid infant and Soluvit supplementation) to the preterm infant

   Or
2. SMOFlipid, (soybean oil, medium chain triglycerides, olive oil and fish oil),(with Vitalipid infant and Soluvit supplementation), where the quotient of Omega 6:3 is 2.5:1 in order to mimic the physiologic relation of fatty acids in cord blood from birth, to the preterm infant.

Thus there is one group of infants (n=45) that will receive Omega-3 in the fatty acid supplementation.

The time on parenteral nutrition and the amount of fatty acids given will be according to clinical routines.

The randomization of the patients will be performed by the controller of the study. Randomization will be in blocks with 10 children in each block.

Data collection

After the investigators have received informed consent from the parents/guardians, blood samples 0.2 ml from the child will be taken according to present clinical practice at if possible from cord (2ml) and at days 0, 7, 14, 28 and in postmenstrual weeks 32, 36 and 40. Blood samples from the mothers for Fatty Acids analyses will be taken after birth, day 7 and at gestational weeks 36 and 40. At the same time (except from day 1), breast milk samples are taken. Length in cm, weight in gram and head circumference in cm are measured weekly.

Screening for ROP will be performed, at least once a week, according to clinical routines using a specific protocol.

The investigators intend to analyze the content of phospholipids which can be done on small amounts of blood, is relatively insensitive to short term fluctuations in intake and mirror the composition of many membranes in the body. The analyses will be made using gas-liquid chromatography. The method has a coefficient of variability of 1-3% for the Fatty Acids concerned.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent from parents/guardians;
2. Subject must be below 28 weeks of gestation

Exclusion Criteria:

1. Detectable clinical gross malformation;
2. Known or suspected chromosomal abnormality, genetic disorder, or syn-drome, according to the investigator's opinion;
3. Clinically significant neuropathy, nephropathy, retinopathy, or other micro- or macrovascular disease requiring treatment, according to the investigator's opinion;
4. Any other condition or therapy that, in the investigator's opinion, may pose a risk to the subject or interfere with the subject's ability to be compliant with this protocol or interfere with interpretation of results.
5. Bleeding disorder.

Ages: 23 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2013-03; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Retinopathy of Prematurity | When the retina is fully vascularised,i.e. at approximately 40 postmenstrual weeks.
  We intend to analyze the content of Fatty Acids and correlate to Retinopathy of Prematurity development and interventional treatment. Analyze of phospholipids can be done on small amounts of blood, is relatively insensitive to short term fluctuations in intake and mirror the composition of many membranes in the body. The analyses will be made using gas-liquid chromatography. The method has a coefficient of variability of 1-3% for the Fatty Acids concerned.

SECONDARY OUTCOMES:
Brain Growth | At 40 postmenstrual weeks and at 2.5 and 6 years.
  Cranial ultrasound will be performed according to clinical praxis. MRI of the brain will be performed at 40 weeks postmenstrual age (PMA) and correlated to interventional treatment.
Length in cm | At 40 postmenstrual weeks and at 2.5 and 6 years.
  Length in cm given in absolute values and in standard deviation scores, at 40 weeks postmenstrual age (PMA) and at 2.5 and 6 years will be correlated to interventional treatment.
Weight in gram | At 40 postmenstrual weeks and at 2.5 and 6 years.
  Weight in gram given in absolute values and in standard deviation scores, at 40 weeks postmenstrual age (PMA) and at 2.5 and 6 years will be correlated to interventional treatment.
Head circumference in cm | At 40 postmenstrual weeks and at 2.5 and 6 years.
  Head circumference in cm given in absolute values and in standard deviation scores, at 40 weeks postmenstrual age (PMA) and at 2.5 and 6 years will be correlated to interventional treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carola Pfeiffer-Mosesson, RN, Principal Investigator — The Queen Silvia Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Cakir B, Hellstrom W, Tomita Y, Fu Z, Liegl R, Winberg A, Hansen-Pupp I, Ley D, Hellstrom A, Lofqvist C, Smith LE. IGF1, serum glucose, and retinopathy of prematurity in extremely preterm infants. JCI Insight. 2020 Oct 2;5(19):e140363. doi: 10.1172/jci.insight.140363. PMID 33004691
- [Derived] Nilsson AK, Pedersen A, Malmodin D, Lund AM, Hellgren G, Lofqvist C, Pupp IH, Hellstrom A. Serum choline in extremely preterm infants declines with increasing parenteral nutrition. Eur J Nutr. 2021 Mar;60(2):1081-1089. doi: 10.1007/s00394-020-02312-2. Epub 2020 Jun 25. PMID 32588218
- [Derived] Lundgren P, Hellgren G, Pivodic A, Savman K, Smith LEH, Hellstrom A. Erythropoietin serum levels, versus anaemia as risk factors for severe retinopathy of prematurity. Pediatr Res. 2019 Aug;86(2):276-282. doi: 10.1038/s41390-018-0186-6. Epub 2018 Sep 18. PMID 30297879
- [Derived] Lofqvist CA, Najm S, Hellgren G, Engstrom E, Savman K, Nilsson AK, Andersson MX, Hard AL, Smith LEH, Hellstrom A. Association of Retinopathy of Prematurity With Low Levels of Arachidonic Acid: A Secondary Analysis of a Randomized Clinical Trial. JAMA Ophthalmol. 2018 Mar 1;136(3):271-277. doi: 10.1001/jamaophthalmol.2017.6658. PMID 29423508
- See also: Homepage — http://www.rop.gu.se